CLINICAL TRIAL: NCT04293640
Title: Neural Respiratory Drive in Pulmonary Hypertension
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Golden Jubilee National Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: 18/CARD/32
Record Dates: First submitted 2020-02-20; First posted 2020-03-03 (Actual); Last update posted 2020-03-03 (Actual); Status verified 2020-03

CONDITIONS: Pulmonary Hypertension
MeSH Terms: conditions — Hypertension, Pulmonary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Parasternal electromyogram measurement — Three electrodes are applied to the chest (two to parasternal muscles, one reference electrode to clavicle). Measurements of EMG signals are recorded on appropriate software.

SUMMARY:
Investigating neural respiratory drive by examining parasternal EMG measurements in patients presenting for assessment of presumed pulmonary hypertension.

DETAILED DESCRIPTION:
NRD can be assessed by measuring parasternal electromyogram (EMG). Readings are taken by applying two small electrodes in the second intercostal space either side of the sternum and one to the shoulder. The electrodes are similar to those used in ECG acquisition. Measurements are then taken during normal breathing and also during maximal breathing effort ('sniff' procedure). Tests may be taken with patient recumbent at 45 degrees and supine. The test is non-invasive, has been safely performed in patients in previous studies and is not anticipated to cause any harm or distress. The total time for measurements will be around 20 minutes per patient.

NRD will be calculated as root mean square of normal tidal breathing as a proportion of maximal inspiratory effort (maximum inspiration from functional reserve capacity, taken as a sniff manoeuvre). Measurements will be performed in a ward based setting at the patient's bedside.

At the end of the inpatient stay for diagnosis, some patients are commenced on treatment and followed up in clinic. It would be the intention of the investigators to reassess these patients at clinic to test NRD and compare how this changes over time compared to other clinical parameters.

In addition, we will collect further readings of NRD in these patients when they attend for their standard follow up appointment. For the majority of patients, this will be after 3-4 months. For a subset of patients with chronic thromboembolic pulmonary hypertension, this may be up to one year after initial readings because these patients may be suitable for surgical intervention, which is not done locally and usually takes place 6-12 months after diagnosis at SPVU.

As such, the investigators intend that a patient will take part in the study for 52 weeks maximum, with most patients taking part for 16 weeks, and the study will not require them to have any additional attendances at hospital outwith their standard hospital admission for diagnosis and clinic follow up.

ELIGIBILITY:
Inclusion Criteria:

* Able to give informed consent
* Being investigated for pulmonary hypertension

Exclusion Criteria:

* Patient is pregnant
* Patient has a diagnosed neuromuscular disorder

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting to Scottish Pulmonary Vascular Unit for investigation of pulmonary hypertension.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2019-02-01 (Actual); Primary Completion 2021-01 (Estimated); Study Completion 2021-01 (Estimated)

PRIMARY OUTCOMES:
Change in neural respiratory drive | 3 months
  Electromyogram (EMG) signals during tidal breathing as a proportion of EMG signals from maximal manoeuvre. Measured at baseline and again 3 months after commencing treatment.

SECONDARY OUTCOMES:
Cross sectional assessment of neural respiratory drive | Baseline test
  Novel data on levels of respiratory drive from parasternal EMG signals in patients with pulmonary hypertension

CONTACTS AND LOCATIONS:
Overall Officials: Martin Johnson, Principal Investigator — NHS Greater Glasgow and Clyde
Locations (1):
- Golden Jubilee National Hospital, Glasgow, United Kingdom

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol (2019-01-19): https://cdn.clinicaltrials.gov/large-docs/40/NCT04293640/Prot_000.pdf
  • Informed Consent Form (2019-01-19): https://cdn.clinicaltrials.gov/large-docs/40/NCT04293640/ICF_001.pdf